CLINICAL TRIAL: NCT03119987
Title: Efficacy of Red Cell Distribution Width as a Predictor of High Risk and Early Mortality in Upper Gastro-intestinal Bleeding
Brief Title: Predictive Role of Red Cell Distribution Width in Upper GI Bleeding Patients
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Other Study IDs: RDWUGI
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Red cell Distribution Width; Risk; Mortality; Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UGIB: Those who was diagnosed as UGI bleeding at emergency department during the study periods. Red cell distribution widths wers checked at all patients.
  Interventions: Diagnostic Test: Red cell distribution widths

INTERVENTIONS:
Diagnostic Test: Red cell distribution widths — Measured value of Red cell distribution widths in initial laboratory result of blood cell counts at emergency department

SUMMARY:
Acute upper-gastrointestinal bleeding (UGIB) is a commonly encountered cause of admission in emergency department (ED). Early risk stratification allows appropriate therapy that may be helpful to advance the patient's morbidity and mortality. Investigators hypothesized that early RDW levels may have an independent, linear relationship with recurrent or massive bleeding in UGIB patients.

DETAILED DESCRIPTION:
This is a retrospective clinical study including the UGI patients in ED. All data will be collected through the electrical medical records. The major endpoints are the high risk patients and 30-days mortality which defined cases of including any of one among the death, re-bleeding, and received the intervention (such as blood transfusion, endoscopic therapy and operation).

Investigators assessed the relationship between initial RDW level and high risk patients and 30-days mortality. In addition, investigators compare the dicrimination power for predicting outcomes between the UGIB scoring system and RDW level.

Univariate and multivariate logistic regression testing and a Cox hazard regression model were used to determine the factors associated with outcome variables. In addition, investigators constructed receiver operating characteristic curves, and the areas under the curves and confidence intervals were calculated to compare the discriminatory power for outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Diagnosis as Upper gastrointestinal bleeding
* Check RDW when patients visited at emergency department

Exclusion Criteria:

* Paediatrics
* Follow up loss
* Data could not be acquired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who visited to emergency department due to Upper gastrointestinal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
High risk | 30 days
  Case of the death or re-bleeding, or blood transfusion or endoscopic therapy or operation.

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, MD, Principal Investigator — Department of Emergency Medicine, Konkuk University School of medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blatchford O, Murray WR, Blatchford M. A risk score to predict need for treatment for upper-gastrointestinal haemorrhage. Lancet. 2000 Oct 14;356(9238):1318-21. doi: 10.1016/S0140-6736(00)02816-6. PMID 11073021
- [Background] van Kimmenade RR, Mohammed AA, Uthamalingam S, van der Meer P, Felker GM, Januzzi JL Jr. Red blood cell distribution width and 1-year mortality in acute heart failure. Eur J Heart Fail. 2010 Feb;12(2):129-36. doi: 10.1093/eurjhf/hfp179. Epub 2009 Dec 20. PMID 20026456
- [Background] Masaoka T, Suzuki H, Hori S, Aikawa N, Hibi T. Blatchford scoring system is a useful scoring system for detecting patients with upper gastrointestinal bleeding who do not need endoscopic intervention. J Gastroenterol Hepatol. 2007 Sep;22(9):1404-8. doi: 10.1111/j.1440-1746.2006.04762.x. PMID 17716345
- [Background] Stanley AJ, Ashley D, Dalton HR, Mowat C, Gaya DR, Thompson E, Warshow U, Groome M, Cahill A, Benson G, Blatchford O, Murray W. Outpatient management of patients with low-risk upper-gastrointestinal haemorrhage: multicentre validation and prospective evaluation. Lancet. 2009 Jan 3;373(9657):42-7. doi: 10.1016/S0140-6736(08)61769-9. Epub 2008 Dec 16. PMID 19091393